CLINICAL TRIAL: NCT01945606
Title: A Single Blind, Placebo Controlled Pilot Study to Explore the Safety and Tolerability of a Single Oral Dose of 30 mg BAY1067197 in Patients With Chronic Heart Failure on the Background of Preexisting Beta-blocker Therapy
Brief Title: Study to Assess the Safety of BAY1067197 in Stable Heart Failure Patients on Standard Therapy Including ß-blocker
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 16718; 2013-001287-34 (EudraCT Number)
Record Dates: First submitted 2013-09-16; First posted 2013-09-18 (Estimated); Last update posted 2019-09-19 (Actual); Status verified 2019-09

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- Placebo and BAY1067197 (Experimental): Patients will get both treatment 1 and 2
  Interventions: Drug: Placebo (treatment 1); Drug: BAY1067197 (treatment 2)

INTERVENTIONS:
Drug: Placebo (treatment 1) — Oral administration of placebo tablets
Drug: BAY1067197 (treatment 2) — Oral administration of a single dose of 30 mg (3×10 mg Tablet) BAY1067197

SUMMARY:
This is a study to investigate the safety and tolerability of the partial A1 agonist BAY1067197 in patients with chronic heart failure. BAY1067197 will be applied as a single dose of 30 mg in addition to standard therapy including a beta-blocker. The aim of the study is to assess if a single oral dose of 30 mg BAY1067197 is well tolerated when given on top of standard therapy for heart failure, particularly ß-blocker treatment.

ELIGIBILITY:
Inclusion Criteria:

* Stable systolic heart failure (heart failure with reduced ejection fraction, heart failure with reduced ejection fraction [HFrEF]; New York Heart Association [NYHA] I-III) in sinus rhythm with a documented ejection fraction (EF) ≤45% within the last 3 months
* Stable standard heart failure (HF) therapy including intermediate to high dose β-blocker with either ≥ 95 mg metoprolol succinate (controlled release tablet), ≥ 5mg Bisoprolol (immediate release [IR] -tablet) or ≥5mg Nebivolol (IR tablet) for at least 4 weeks. Additional intake of angiotensin-converting enzyme (ACE) inhibitors or angiotensin receptor blockers and optional aldosterone-receptor antagonists, diuretics or digitalis is allowed
* Men or confirmed postmenopausal women (defined as being amenorrheic for longer than 2 years with an appropriate clinical profile, e.g. age appropriate and a history of vasomotor symptoms) or women without childbearing potential based on surgical treatment such as bilateral tubal ligation, bilateral ovarectomy, or hysterectomy (documented by medical report verification). Men enrolled in this study must agree to use adequate barrier birth control measures during the treatment period of the study and for 12 weeks after receiving the investigational medicinal product (IMP)
* Male patients must agree not to act as sperm donor for 12 weeks after dosing
* Ethnicity: White
* Body mass index (BMI): above/equal 18.0 and below/equal 29.9 kg/m²
* Age: 18 to 75 years (inclusive) at the first screening visit

Exclusion Criteria:

* Biventricular pacing/active cardiac resynchronization therapy (CRT) device
* Dependency on pacemaker or implantable cardioverter-defibrillator (ICD) device with pacemaker dependency (a paced ventricular rhythm > 5% of heart activity)
* A history of relevant diseases of vital organs other than the heart, of the central nervous system or other organs
* Known hypersensitivity to the study preparations (active substances or excipients of the preparations) or to any other β-blocker
* Current or history of AV-Block > I°
* Unstable condition, indicated by requirement of IV drug (diuretic, inotrope, etc.) or NYHA IV
* Acute Coronary Syndrome (defined as unstable angina [UA], non-ST elevation myocardial infarction [NSTEMI], ST elevation myocardial infarction [STEMI]) within 3 months prior to first study drug administration
* History of asthma or chronic obstructive pulmonary disease (COPD) ≥ global initiative for chronic obstructive lung disease (GOLD) II and/or allergic asthma
* Women of childbearing potential, pregnancy or breastfeeding

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2013-11-29 (Actual); Primary Completion 2014-09-09 (Actual); Study Completion 2015-03-17 (Actual)

PRIMARY OUTCOMES:
Number of patients with occurrence of AV-Block > I° | up to 48 hours

SECONDARY OUTCOMES:
Pharmacokinetic profile determined by tmax | up to 24 hours
Pharmacokinetic profile determined by t1/2 | up to 22 days
Heart rate | multiple time points up to 24 hours
Blood pressure | multiple time points up to 24 hours
Number of participants with adverse events as a measure of safety and tolerability | up to 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Groningen, Netherlands

REFERENCES:
- See also: Click here to find results for studies related to Bayer products — http://clinicaltrials.bayer.com/